CLINICAL TRIAL: NCT03980561
Title: Varenicline for the Treatment of DSM 5 Cannabis Use Disorder in Adults
Brief Title: UH3 Varenicline for Cannabis Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00089933
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Cannabis Use Disorder
Keywords: marijuana; substance use
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline (Experimental): 2 mg daily
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): 2 mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Active medication
  Other Names: Chantix, Apo-Varenicline
  Arms: Varenicline
Drug: Placebo — Inactive medication
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Marijuana is the most commonly used illicit drug. There is high demand for effective interventions for cannabis use disorder, yet few specific treatments for have been developed. This study will evaluate the efficacy of varenicline for reducing marijuana use in people who use marijuana frequently.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-5 criteria for cannabis use disorder and use cannabis at least 3 days per week in the last 30 days.
* Express interest in receiving treatment for cannabis use disorder and reducing use.
* Must be at least 18 years of age.
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial.
* Must consent to random assignment, and be willing to commit to medication ingestion.
* Must be able to read and provide informed consent.
* Must have body weight >110lbs (50kg) and have BMI between 18 and 35kg/m2
* Must function at an intellectual level and have knowledge of the English language to sufficiently allow for accurate completion of assessments.

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study.
* Individuals with severe renal impairment (creatinine clearance less than 30 mL per minute).
* Lifetime history of DSM-5 Bipolar I or II Disorder, Schizophrenia or other psychotic disorder. Stably treated MDD, Dysthymia, GAD, Social Phobia, and Specific Phobia diagnoses are acceptable (i.e. same dose of medication has been prescribed for at least 2 months prior to screening and no changes in current medication expected during course of the trial).
* Past year or current posttraumatic stress disorder.
* Subjects who are actively suicidal, or who report suicidal ideation (SI) with intent or plan in the past year.
* Subjects who have a SBQ R total score ≥8, or for whom the investigator judges that a risk assessment by a qualified medical professional is required. Subjects answering 'yes' on questions 4 or 5 of C-SSRS will be referred to assessment by a qualified mental health professional.
* Suicidal behavior within the past 10 years or a lifetime history of serious or recurrent suicidal behavior.
* Concomitant use of psychotropic medications, with the exception of stable doses (defined as no dosing adjustments in the past two months) of non-MAO-I antidepressants, non-benzodiazepine anxiolytics, and ADHD medications.
* Current use of medications prescribed for mania or psychosis.
* Current use of buproprion or nortryptiline.
* Moderate or severe non-cannabis substance use disorders within the past 60 days with the exception of tobacco use disorder.
* Past year or current moderate or severe alcohol use disorder.
* Individuals taking an investigational agent within the last 30 days before baseline visit.
* Individuals with clinically significant medical disorders or lab abnormalities.
* Any individual at screening with SGOT (AST) or SGPT (ALT) greater than 3 times the upper limit of normal and/or total bilirubin greater than two times the upper limit of normal.
* Individuals with clinically significant cardiovascular disease in the past 6 months (e.g., myocardial infarction, CABG, PTCA, severe or unstable angina, serious arrhythmia, or any clinically significant ECG conduction abnormality.
* Individuals with clinically significant cerebrovascular disease in the past 6 months such as TIA, CVA, or stroke.
* Hypersensitivity to varenicline.
* Individuals who have participated in the clinical trial of any investigative compound within the last 60 days
* Individuals who are on probation or under a mandate to obtain treatment.
* Individuals with plans to initiate or change frequency of attendance at self-help meetings (e.g. AA, NA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 90 | 84
Completed | 61 | 59
Not Completed | 29 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 90 | 84 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 84 | 173
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 57 | 58 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 84 | 72 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 28 | 53
  White | 57 | 50 | 107
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 90 | 84 | 174

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Varenicline vs. Placebo for Reducing Total Number of Weekly Cannabis Use Sessions
Description: Cannabis use reduction was measured by daily substance use logs/self-report and examined as the total number of use sessions reported at each weekly visit.
Time Frame: Treatment phase Weeks 6-12
Population: Week 6 participants
Measure: Mean (Standard Deviation); unit: number of weekly use sessions
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 68 | 63
number of weekly use sessions
  Week 6 | 10.3 (8.2) | 11.6 (11.4)
  Week 7: number analyzed (Participants) | 62 | 60
  Week 7 | 9.4 (8.2) | 11.7 (11.4)
  Week 8: number analyzed (Participants) | 63 | 59
  Week 8 | 9.4 (7.9) | 10.5 (11.3)
  Week 9: number analyzed (Participants) | 62 | 57
  Week 9 | 8.5 (7.6) | 9.7 (10.2)
  Week 10: number analyzed (Participants) | 58 | 55
  Week 10 | 9.2 (7.7) | 10.7 (10.8)
  Week 11: number analyzed (Participants) | 54 | 54
  Week 11 | 8.4 (7.5) | 11.8 (12.8)
  Week 12: number analyzed (Participants) | 57 | 56
  Week 12 | 8.4 (8.6) | 11.5 (11.1)

2. Secondary Outcome: Safety and Tolerability of Varenicline vs. Placebo When Used for Cannabis Use Disorder
Description: Comparing the frequency of participant-reported treatment-emergent AEs between treatment groups. Of particular interest will be AEs leading to medication discontinuation and the occurrence of treatment-related serious AEs.
Time Frame: 12 weeks (across the active treatment period)
Population: Participants reporting an adverse event during 12 week active treatment period
Measure: Number; unit: number of adverse events
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 81 | 70
number of adverse events
  All reported adverse events | 406 | 300
  Medication-related adverse events: number analyzed (Participants) | 75 | 47
  Medication-related adverse events | 238 | 115
  Serious adverse events related to treatment: number analyzed (Participants) | 1 | 0
  Serious adverse events related to treatment | 0 |
  Adverse events resulting in temporary or permanent medication discontinuation: number analyzed (Participants) | 11 | 9
  Adverse events resulting in temporary or permanent medication discontinuation | 26 | 14

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of consent through last study visit (approximately 14 weeks).
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/90 | 0/84
Other Adverse Events (participants affected / at risk) | 81/90 | 70/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=90) | Placebo (N=84)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=90) | Placebo (N=84)
anxiety/depression (Psychiatric disorders) | 12 (13) | 15 (17)
decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 11 (11)
dream disturbance (General disorders) | 41 (54) | 21 (32)
fatigue (General disorders) | 7 (7) | 4 (4)
headache (General disorders) | 16 (21) | 25 (28)
insomnia (General disorders) | 24 (24) | 20 (22)
irritability (General disorders) | 11 (13) | 11 (12)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 (10) | 13 (21)
nausea (Gastrointestinal disorders) | 49 (64) | 20 (24)
night sweats (General disorders) | 5 (6) | 5 (6)
other GI (Gastrointestinal disorders) | 25 (45) | 23 (29)
URI/cold symptoms (Infections and infestations) | 20 (23) | 14 (17)
vomiting (Gastrointestinal disorders) | 21 (27) | 9 (10)

LIMITATIONS AND CAVEATS:
Varenicline's efficacy for cannabis use disorder may vary by sex; however, this study was not powered to fully explore potential sex differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03980561/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03980561/ICF_000.pdf